CLINICAL TRIAL: NCT07403630
Title: INTEGRATIVE "MULTI-OMICS" AND FUNCTIONAL PLATFORM FOR THE COMPLETE DIAGNOSTIC CHARACTERIZATION OF TUMORS: THE ITALIAN TUMOR CHEMOGENOMIC PROFILER (IT-TCP)
Acronym: IT-TCP POS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Giovanni Roti, Full Professor, Azienda Ospedaliero-Universitaria di Parma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5756
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Acute Leukemia; Multiple Myeloma; Chronic Myeloproliferative Neoplasm; Squamous Cell Carcinoma; Pleural Mesothelioma; Pancreatic Cancer; Bladder Cancer; Ovarian Cancer; Melanoma; Pediatric Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Multiple Myeloma; Myeloproliferative Disorders; Carcinoma, Squamous Cell; Mesothelioma, Malignant; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Melanoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other)
  Interventions: Other: Peripheral blood and bone marrow withdrawal

INTERVENTIONS:
Other: Peripheral blood and bone marrow withdrawal — Biological characterization of primary samples from patients diagnosed with haematological or solid neoplasms defined as high-risk

SUMMARY:
This pre-clinical, experimental study will involve primary samples from patients diagnosed with haematological or solid neoplasms defined as high-risk.

It will be prospective, based on consecutive enrolment of eligible patients at each participating institution.

DETAILED DESCRIPTION:
This pre-clinical, experimental study will involve primary samples from patients diagnosed with haematological or solid neoplasms defined as high-risk.

It will be prospective, based on consecutive enrolment of eligible patients at each participating institution. Patients will be enrolled based on their biological and clinical characteristics at the time of diagnosis. This will include patients with metastatic disease, as well as those with recurrent or refractory disease, particularly where the therapeutic indication is not supported by internationally recognised guidelines.

ELIGIBILITY:
Inclusion criteria:

Patients aged one year and over who are referred to the centres involved in the protocol (Azienda Ospedaliero-Universitaria di Parma, University of Parma, University of Perugia and Azienda Ospedali Riuniti Villa Sofia-Cervello of Palermo).

* Patients with an established diagnosis of haematological or solid organ malignancy, including haematological or solid malignancies characteristic of the paediatric age group.
* Patients diagnosed with relapsed, refractory and/or metastatic haematological or solid malignancy. Patients may be enrolled regardless of the extent and type of previous therapy. Patients may also be enrolled if they are undergoing active treatment at the time of evaluation.

Patients must have the capacity to understand the investigative nature of the study and provide informed consent in writing. For patients under the age of 12 years, consent will be provided by the parent/legal guardian according to international guidelines. For patients aged 12 to 17 years, consent will be provided by the patient and the parent/legal guardian according to the mature minor principle.

Exclusion criteria:

* Patients younger than 1 year old
* Patients with active, uncontrolled infections

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-02-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the rate of change in therapeutic indication of disease from standard-of-care. | At baseline

SECONDARY OUTCOMES:
Evaluation of the possible use of the IT-TCP platform on the clinical level | At baseline
Creation of an IT platform to store and manage the data generated | At baseline

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - AO Riuniti Villa Sofia-Cervello di Palermo, Palermo, Palermo
  - University of Perugia, Perugia, Perugia